CLINICAL TRIAL: NCT04221321
Title: An Open-label, Randomized, Multiple-dose, Replicated Crossover Study to Evaluate Drug-drug Interaction Following Co-administration of Tegoprazan or RAPA114 With Atorvastatin in Healthy Adults
Brief Title: Effect of Tegoprazan or RAPA114 on Pharmacokinetic of Atorvastatin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_114
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-06

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin; tegoprazan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atorvastatin 40 mg (Placebo Comparator): Oral administration of Atorvastatin 40 mg tablet once daily for 7 days
  Interventions: Drug: Atorvastatin 40 mg
- Atorvastatin 40 mg + Tegoprazan 50 mg (Experimental): Oral administration of Atorvastatin 40 mg tablet and Tegoprazan 50 mg tablet once daily for 7 days
  Interventions: Drug: Atorvastatin 40 mg; Drug: Tegoprazan 50 mg
- Atorvastatin 40 mg + RAPA114 (Active Comparator): Oral administration of Atorvastatin 40 mg tablet and RAPA114 tablet once daily for 7 days
  Interventions: Drug: Atorvastatin 40 mg; Drug: RAPA114

INTERVENTIONS:
Drug: Atorvastatin 40 mg — Atorvastatin 40 mg
  Other Names: Lipitor
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Atorvastatin 40 mg + Tegoprazan 50 mg
Drug: RAPA114 — RAPA114 tablet
  Arms: Atorvastatin 40 mg + RAPA114

SUMMARY:
This study aims to evaluate the influence of tegoprazan or RAPA114 on the Pharmacokinetic characteristics of atorvastatin following co-administration of tegoprazan or RAPA114 in healthy adult volunteers.

DETAILED DESCRIPTION:
[Pharmacokinetic Assessments] : Blood concentration of atorvastatin, 2-OH atorvastatin

* Primary outcome: AUCτ, Css,max of atorvastatin
* Secondary outcome: Tss,max of atorvastatin, AUCτ, Css,max of 2-OH atorvastatin, metabolic ratio

[Sefety Assessments]

: Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 19 to 55 years (inclusive) at the time of his consent.
* Body mass index (BMI) ≥ 19.0 and ≤ 27.0 kg/m2 at screening.
* Decides to participate voluntarily in the trial after being fully informed of and understanding the study completely, and provides the written informed consent to participate in the trial and to comply with the trial-specific requirements.
* Has the ability and willingness to participate in the entire period of clinical trial.

Exclusion Criteria:

* A subject with clinically significant disease or history of hepatobiliary, renal, gastrointestinal, cardiovascular, musculoskeletal, endocrine, respiratory, neuropsychiatry or hemato-oncologic system, etc.
* A subject with a history of hypersensitivity reactions to main constituents of or identical affiliation of the investigational products (ex, HMG-CoA reductase inhibitor, gastric acid suppressants), or have allergic diseases that require treatment.
* A subject with a history of genetic myopathy or family history.
* A subject who has participated in other clinical trials and received the investigational products within 180 days prior to the randomization.
* A subject who received any medications or foods that could significantly affect the absorption, distribution, metabolism, or excretion of an investigational product within 30 days prior to the randomization.
* A subject with history of whole blood donation within 60 days, or with blood components or received transfusion within 30 days prior to the randomization.
* A subject with continued consumption of alcohol more than 140 g per week.
* A subject with AST, ALT, or γ-GT levels exceeding 1.5 times of the upper limit of the reference range in the screening test.
* A subject with a calculated glomerular filtration rate of less than 60 mL / min / 1.73 m2 in the screening test.
* A subject with any positive result on serology tests for hepatitis B, hepatitis C, HIV or syphilis in the screening test.
* A subject with galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose malabsorption, etc.
* Male subject who don't have willing to accept medically acceptable contraceptive methods during the course of clinical trial, or who plan to provide sperm.
* A subject who is determined to be ineligible to participate in the clinical trial by the investigator for other reasons.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
AUCτ of atorvastatin | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  Area under the plasma drug concentration-time curve at steady state
Css,max of atorvastatin | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  Maximum concentration of drug in plasma of atorvastatin at steady state

SECONDARY OUTCOMES:
Tss,max of atorvastatin | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  Time to Cmax at steady state
AUCτ of 2-OH atorvastatin | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  Area under the plasma drug concentration-time curve at steady state
Css,max of 2-OH atorvastatin | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  Maximum concentration of drug in plasma of 2-OH atorvastatin at steady state
metabolic ratio | Pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in each period
  AUCτ of 2-OH atorvastatin / AUCτ of atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Jung-ryul Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea